CLINICAL TRIAL: NCT05046327
Title: A Multicenter, Open-Label Study to Evaluate the Safety and Efficacy of Avatrombopag and Remission Rates in Adults With Immune Thrombocytopenia (ITP) of ≤6 Months Duration
Brief Title: Open-Label Study to Evaluate the Safety and Efficacy of Avatrombopag and Remission Rates in Adults With ITP of ≤6 Months
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Corporate Decision
Sponsor: Sobi, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVA-ITP-306
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — avatrombopag; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 20 mg Avatrombopag daily (Experimental): Avatrombopag
  Interventions: Drug: Avatrombopag 20 mg Oral Tablet

INTERVENTIONS:
Drug: Avatrombopag 20 mg Oral Tablet — Avatrombopag administered at a frequency to maintain a target platelet count between ≥50 and ≤150×10⁹/L
  Other Names: Doptelet

SUMMARY:
This study will evaluate the safety and efficacy of avatrombopag in subjects with a confirmed diagnosis of primary ITP (≤6 months duration) over 26 weeks of treatment, and also evaluate the incidence of ITP remission.

DETAILED DESCRIPTION:
This phase 3b, multi-center, open-label study will enroll approximately 75 adult subjects with a confirmed diagnoses of primary ITP (≤6 months duration) who have had a previous response to a first line treatment. The study will consist of a 26-week treatment period to evaluate the safety and efficacy of avatrombopag. Subjects with platelet counts ≥50×10⁹/L at Week 26 may enter a dose-tapering period in which the dose of avatrombopag will be decreased for up to 16 weeks until avatrombopag treatment is discontinued and the platelet count is maintained ≥50×10⁹/L. Once avatrombopag treatment has been discontinued, the subjects will enter a remission evaluation period of up to 24 weeks to evaluate whether they have entered a state of remission.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years of age at Screening.
2. Subject must be able to provide informed consent.
3. Subject has a confirmed diagnosis of primary ITP according to the International Consensus Report on the Investigation and Management of Primary ITP within the previous 6 months prior to Visit 1 and has had a previous response to a first line treatment (corticosteroids, IVIg, or anti-D), in the opinion of the Investigator.
4. Subject has at least one platelet count <30×10⁹/L at any time during the screening period or at the Baseline visit.
5. Females of childbearing potential must have a negative pregnancy test at Screening and Baseline.
6. Female subjects of childbearing potential who are sexually active and male subjects who are sexually active must agree to use effective methods of contraception.
7. Subject is willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

1. Thrombocytopenia due to a known condition other than primary ITP (e.g., systemic lupus erythematosus, H. pylori infection, splenomegaly, chronic liver disease).
2. Any history of arterial or venous thrombosis, including partial or complete thrombosis (history of superficial thrombophlebitis is not exclusionary).
3. Subjects with known inherited thrombocytopenia (e.g., MYH-9 disorders).
4. History of myelodysplastic syndrome (MDS) or other hematologic malignancies.
5. Current history of significant cardiac arrhythmias or decompensated congestive heart failure.
6. History of hepatitis B (HBV), hepatitis C (HCV), or human immunodeficiency virus (HIV).
7. Previous use of eltrombopag, romiplostim, recombinant human TPO or other platelet-producing agents.
8. Surgical resection of the spleen.
9. Previous use of mycophenolate mofetil (MMF), rituximab (or other B-cell lymphocyte depleting agents), mercaptopurine (6-MP) or alkylating agents.
10. Concurrent malignant disease, other than non-melanoma skin cancer or cervical cancer in-situ.
11. Known allergy to avatrombopag or any of its excipients.
12. Subject is unable to take oral medication or has a malabsorption syndrome or any other uncontrolled gastrointestinal condition.
13. Enrollment in another clinical study with any investigational drug or device within 30 days of Day 1/Visit 2 (or 5 half-lives, whichever is longer); however, participation in observational studies is permitted.
14. Any clinically relevant abnormality which makes the subject unsuitable for participation in the study, in the opinion of the Investigator.
15. Considered unable or unwilling to comply with the study protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-14 (Estimated); Primary Completion 2024-04-06 (Estimated); Study Completion 2025-02-19 (Estimated)

PRIMARY OUTCOMES:
Cumulative Number of Weeks of Platelet Response | 6 Months of Active Treatment
  Cumulative number of weeks of platelet response in which the platelet count is ≥50×10⁹/L during 6 months of treatment in the absence of rescue therapy.

SECONDARY OUTCOMES:
Durable Platelet Response | 8 Weeks of Treatment
  Durable platelet response as defined by the incidence of subjects who have at least 6 out of 8 weekly platelet counts ≥50×10⁹/L during the last 8 weeks of treatment.
Incidence of ITP remission | 24 Consecutive Weeks
  Incidence of ITP remission as defined by platelet count ≥50×10⁹/L for 24 consecutive weeks with no ITP treatments (concomitant or rescue).
Incidence of subjects achieving a platelet count response | 6 Months of Active Treatment
  Incidence of subjects achieving a platelet count response (≥50×10⁹/L) during the active treatment period of the study.

IPD SHARING:
Plan to Share IPD: No